CLINICAL TRIAL: NCT01712607
Title: Preoperative Warm-up in Gynecologic Surgery Using a Virtual Reality Simulator.
Brief Title: Preoperative Warm-up in Gynecologic Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephan Polterauer, MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Warm-Up-1.0
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Gynecologic Disorders
Keywords: laparoscopy; surgery; warm-up; preoperative; surgical skills
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm-Up (Experimental): Surgery after warm-up task Preoperative Warm-Up training
  Interventions: Other: Preoperative Warm-Up training
- No Warm-up (No Intervention): Surgery without warm-up exercise

INTERVENTIONS:
Other: Preoperative Warm-Up training — Preoperative Warm-Up training
  Arms: Warm-Up

SUMMARY:
Background and Objectives: All modern surgical procedures require a high level of cognitive and psychomotor skills achieved using different training methods, but could be influenced by fatigue and other psychological factors. We evaluate the effect of warm-up exercises on operative laparoscopic performances in gynecologic laparoscopic procedures.

Methods: The surgical team operates on a consecutive series of 20 patients and perform laparoscopic salpingo-oophorectomy. Patients are randomly allocated in 2 groups: group A to be operated on without warm-up exercises and group B to be operated on after a short-term warm-up. All patients are operated on by the same surgical team. The full-time records of the operation were analyzed by 2 independent reviewers. Laparoscopic procedures are recorded and assessed by 2 independent observers using the generic OSATS rating scale. A training module using the Lap Sim simulator was designed for the warm-up.

ELIGIBILITY:
Inclusion Criteria:

* residents or faculty at the Dept. of Gynecology and Obstetrics
* completed skills training

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Surgical performance | During surgery
  Surgical Performance will be assessed using Objective structured assessment of technical skills (OSATS)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Polterauer, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. Gynecology and Obstetrics, Medical University of Vienna, Austria, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Polterauer S, Husslein H, Kranawetter M, Schwameis R, Reinthaller A, Heinze G, Grimm C. Effect of Preoperative Warm-up Exercise Before Laparoscopic Gynecological Surgery: A Randomized Trial. J Surg Educ. 2016 May-Jun;73(3):429-32. doi: 10.1016/j.jsurg.2015.11.017. Epub 2016 Jan 14. PMID 26778744
- See also: Surgical Skills Training Center, Medical University of Vienna — http://www.meduniwien.ac.at/SSTC/